CLINICAL TRIAL: NCT01094483
Title: A Phase I Prospective, Randomized, Double-blind, Placebo-controlled Study Assessing Inhibition of Serum Thromboxane B2 Levels With PN 400 and Low Dose Aspirin
Brief Title: A Study Assessing Inhibition of Serum Thromboxane B2 Levels With PN400 and Low Dose Aspirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: POZEN (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D1120C00036
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Platelet Inhibition
Keywords: Thromboxane B2
MeSH Terms: interventions — acetylsalicylic acid lysinate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): PN400 + ASA
  Interventions: Drug: PN400; Drug: ASA
- 2 (Placebo Comparator): Placebo + ASA
  Interventions: Drug: ASA; Drug: Placebo

INTERVENTIONS:
Drug: PN400 — naproxen 500 mg/esomeprazole 20 mg oral tablet
  Arms: 1
Drug: ASA — Asprin 81 mg enteric coated tablet
  Other Names: Asprin
Drug: Placebo
  Arms: 2

SUMMARY:
The primary hypothesis of this study is that concomitant multiple-dose administration of PN 400 does not interfere with the platelet inhibitory effects of enteric-coated low-dose aspirin (81 mg), as measured by serum thromboxane B2 inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Stable without clinically significant disease

Exclusion Criteria:

* Use of NSAID within 2 weeks
* Type 1 or 2 DM
* GI disorder

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic: Mean percent inhibition of serum thromboxane B2 | measured on the morning of Day 6 (Period 1), and 24 hours after the Day 10 morning dose of aspirin (ie, Day 11) in Period 2
Safety: Parameters include: physical examination, vital signs, clinical laboratory tests, adverse events | during approx 6 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schutz, MD, Principal Investigator — Quintiles Phase 1 Services; Catherine Datto, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Angiolillo DJ, Hwang C, Datto C, Desai B, Sostek M. Impact of a fixed-dose combination of naproxen and esomeprazole magnesium on serum thromboxane B2 inhibition by low-dose aspirin over 5 days in healthy adults: a phase I, randomized, double-blind, placebo-controlled, noninferiority trial. Clin Ther. 2011 Dec;33(12):1883-93. doi: 10.1016/j.clinthera.2011.10.009. Epub 2011 Nov 10. PMID 22078153